CLINICAL TRIAL: NCT07353710
Title: A Study on the Acquisition of 2D ICE Images With the CHORUS IDx System in Subjects Undergoing an Ablation Procedure
Acronym: SONAR-ICE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PF339
Record Dates: First submitted 2025-12-12; First posted 2026-01-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Atrial Arrhythmia; Intracardiac Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Subjects with at least one ICE image collected with the investigational system
  Interventions: Device: ICE Image Acquisition

INTERVENTIONS:
Device: ICE Image Acquisition — ICE image acquisition using the investigational device

SUMMARY:
A first-in-human prospective data collection study including subjects who are planned to undergo an ablation procedure for any atrial arrhythmia as per medical judgement and the site's standard practice, represents the most viable means to collect human anatomy ICE images for the purpose of software development.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able and willing to provide written informed consent prior to any study procedure.
2. Subjects who are planned for an ablation procedure for any atrial arrhythmia using any commercially available Boston Scientific Ablation System, per physician's judgement and hospitals' standard practice.
3. Subjects who are willing and able to participate in all testing and assessments associated with this clinical study at an approved clinical investigation center.
4. Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Any of the following cardiac implanted devices

   * Any prosthetic mitral or tricuspid heart valve, such as ring, repairs or clips
   * Atrial septal defect (ASD) occluders including interatrial baffle, closure device, patch, or patent foramen ovale or ASD occluder
2. Subjects with contraindications related to the use of the CHORUS IDx™ System:

   * Subjects with inadequate vascular access
   * Subjects with active systemic infection
   * Subjects with presence of a known intracardiac thrombus in the chamber of use
3. Women who are confirmed to be pregnant or lactating at the time of the Index Procedure
4. Presence of other medical conditions, that, in the investigator's opinion, could limit the subject's ability to participate in the study
5. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the Sponsor to determine eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of procedure related serious adverse events and all adverse events | 7 Days
  Incidence of safety events that have occurred in subjects in whom the investigational device has been inserted, including:
  * Index Procedure related serious adverse events up to day 7 after the Index Procedure
  * All adverse events
  Note: Imaging data will be used for development and validation of the software.

IPD SHARING:
Plan to Share IPD: No